CLINICAL TRIAL: NCT04147455
Title: Preventing Sexual Violence in College Men: Adaptation and Impact Evaluation of RealConsent for Use in Vietnam
Brief Title: Preventing Sexual Violence in College Men: RealConsent for Use in Vietnam
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Center for Creative Initiatives in Health and Population (Other)
Responsible Party: Principal Investigator, Kathryn Yount, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00099860
Record Dates: First submitted 2019-10-30; First posted 2019-11-01 (Actual); Results first posted 2021-07-14 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-09

CONDITIONS: Sexual Violence
Keywords: Behavioral intervention; Violent behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RealConsent (Experimental): Participants randomized to this study arm will receive an adapted program of RealConsent.
  Interventions: Behavioral: Adapted RealConsent
- Health Education Control Condition (Active Comparator): Participants in the control arm will receive a web-based health promotion program.
  Interventions: Behavioral: Health Education Control Condition

INTERVENTIONS:
Behavioral: Adapted RealConsent — The program is a novel, theory-driven, evidence-based serial drama and educational program tailored to young men and delivered in six episodes via the web. Participants will view six 30-minute modules designed to prevent sexual violence in young men
  Arms: RealConsent
Behavioral: Health Education Control Condition — Participants will view six 30-minute web-based serial drama modules designed to promote health.
  Arms: Health Education Control Condition

SUMMARY:
This study is a randomized controlled trial using a web-based adaptation of the RealConsent program among eligible college men in Hanoi, Vietnam. This study will test the impact of the program on promoting prosocial bystander behavior and preventing sexual violence perpetration, through improvements in the seven knowledge, attitudinal, and emotional mediators over a seven month study period, with a baseline survey and two follow-up surveys.

DETAILED DESCRIPTION:
Sexual violence is any sexual act committed against a person without freely given consent. Men and women may experience sexual violence, but most victims are women. Women's first experiences of sexual violence often occur in adolescence. In Asia and the Pacific, about 14% of sexually experienced adolescent girls report forced sexual debut. Thus, early prevention with men is critical; yet, young men often are difficult to reach and may resist programs that target sexual violence, not seeing themselves as potential perpetrators. Prevention with men that integrates a bystander framework, which treats men as "allies" of women, is one way to target attitudes and behaviors while decreasing resistance to participation. In this study, the researchers will adapt an existing program for use with men attending one of two universities in Hanoi, Vietnam. This study will test the impact of the adapted program on knowledge/attitudinal/emotional mediators, and in turn, on sexual violence perpetration and prosocial bystander behavior in this target group. The adapted program is a novel, six-session, web-based serial drama and educational program designed to prevent sexual violence perpetration and to enhance prosocial bystander behavior in young men. The program has reduced the incidence of sexual violence among men attending an urban, public university in the Southeastern United States.

After conducting interviews with men and women, and focus group discussions with college men and university stakeholders the researchers will produce a web-based adaptation of the RealConsent program in Vietnam. The researchers will then conduct a randomized controlled trial to test the impact of the adapted program, relative to a health-education control condition, on knowledge/attitudinal/emotional mediators, and in turn, on sexually violent behaviors, and prosocial bystander behavior in freshmen men attending two universities in Hanoi. This project will be the first to adapt and to test the impact of a novel, theoretically grounded, web-based intervention to prevent sexual violence perpetration and to promote prosocial bystander behavior among young men for use in a middle-income country. If this study shows that the adapted program is effective cross-culturally, it will have exceptional potential for scale-up to prevent men's perpetration of sexual violence against women globally.

ELIGIBILITY:
Inclusion Criteria:

* Identifying as heterosexual or bisexual
* Enrolled as a freshman at Hanoi Medical University or Thang Long University on 9/1/2019

Exclusion Criteria:

* None

Ages: 18 Years to 24 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 793 (Actual)
Dates: Start 2019-09-11 (Actual); Primary Completion 2020-12-02 (Actual); Study Completion 2020-12-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Yount, PhD, Principal Investigator — Emory University
Locations (2):
- Vietnam (2):
  - Thang Long University, Hanoi
  - Hanoi Medical University, Hanoi

IPD SHARING:
Plan to Share IPD: Yes
All de-identified data will be available for sharing, including data dictionaries, with the exception of potentially sensitive items on sexual violence perpetration.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will be made available for sharing beginning 12 months after the end of the study, with no end date.
Access Criteria: Data are available for sharing with researchers requesting data from the Principal Investigator and study steam, providing the analysis plan and study aims are approved. Data will be shared via a secure link through Emory Box as STATA, Excel, and SAS files.

REFERENCES:
- [Background] Yount KM, Minh TH, Trang QT, Cheong YF, Bergenfeld I, Sales JM. Preventing sexual violence in college men: a randomized-controlled trial of GlobalConsent. BMC Public Health. 2020 Sep 1;20(1):1331. doi: 10.1186/s12889-020-09454-2. PMID 32873262
- [Derived] Yount KM, Cheong YF, Bergenfeld I, Trang QT, Sales JM, Li Y, Minh TH. Impacts of GlobalConsent, a Web-Based Social Norms Edutainment Program, on Sexually Violent Behavior and Bystander Behavior Among University Men in Vietnam: Randomized Controlled Trial. JMIR Public Health Surveill. 2023 Jan 27;9:e35116. doi: 10.2196/35116. PMID 36705965

RESULTS

PARTICIPANT FLOW:
Groups:
- Health Education Control Condition: Participants in the control arm received a health promotion program where they watched six 30-minute web-based serial drama modules designed to promote health.
- RealConsent: Participants randomized to this study arm received the adapted program of RealConsent. The RealConsent program is a novel, theory-driven, evidence-based serial drama and educational program tailored to young men and delivered in six episodes via the web. Participants viewed six 30-minute modules designed to prevent sexual violence in young men.
Period: Overall Study
Arm/Group | Health Education Control Condition | RealConsent
Started | 397 | 396
Completed | 375 | 364
Not Completed | 22 | 32

BASELINE CHARACTERISTICS:
Population: Participants were first-year male students matriculating into one of two universities in Hanoi, Vietnam.
Groups:
- Total: Total of all reporting groups
Arm/Group | Health Education Control Condition | RealConsent | Total
Number analyzed (Participants) | 397 | 396 | 793
Age, Continuous [Mean (Standard Deviation); unit: years] | 18.06 (0.32) | 18.07 (0.44) | 18.06 (0.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 397 | 396 | 793
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 397 | 396 | 793
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Vietnam | 397 | 396 | 793

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Contact Sexual Violence Via Physical Tactics
Description: Acts of contact sexual violence using physical tactics (force or threat of harm) were assessed using 7 items from the Sexual Experiences Survey. The 7 items are scored on a scale from 0 (zero acts) to 3 (multiple acts), indicating how many times the participant reported engaging in a specific tactic in order to engage in contact sexual violence, including unwanted touching, rape, and attempted rape. The numbers of participants indicating they used physical tactics at least once (scores of 1 or 2) to perpetrate any of seven acts of contact physical violence (in the past twelve months, for the baseline assessment, or since last completing the questionnaire) are presented here.
Time Frame: Baseline, immediately after completing the 3 week intervention, 6 months after completing the intervention
Population: This analysis includes participants who completed the assessments at the indicated time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Health Education Control Condition | RealConsent
Number analyzed (Participants) | 397 | 396
Participants
  Baseline | 23 | 32
  Immediately post-intervention: number analyzed (Participants) | 377 | 374
  Immediately post-intervention | 46 | 35
  6 months post-intervention: number analyzed (Participants) | 375 | 364
  6 months post-intervention | 39 | 31

2. Primary Outcome: Number of Participants Reporting Contact Sexual Violence Via Non-physical Tactics
Description: Acts of contact sexual violence using non-physical tactics (verbal coercion, lying, or intoxication) were assessed using 7 items from the Sexual Experiences Survey. The 7 items are scored on a scale from 0 (zero tactics) to 3 (multiple tactics), indicating how many times the participant reported engaging in a specific tactic in order to engage in contact sexual violence, including unwanted touching, rape, and attempted rape. The numbers of participants indicating they used non-physical tactics at least once (scores of 1 or 2) to perpetrate any of seven acts of contact physical violence (in the past twelve months, for the baseline assessment, or since last completing the questionnaire) are presented here.
Time Frame: Baseline, immediately after completing the 3 week intervention, 6 months after completing the intervention
Population: This analysis includes participants who completed the assessments at the indicated time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Health Education Control Condition | RealConsent
Number analyzed (Participants) | 397 | 396
Participants
  Baseline | 41 | 48
  Immediately post-intervention: number analyzed (Participants) | 377 | 374
  Immediately post-intervention | 65 | 47
  6 months post-intervention: number analyzed (Participants) | 375 | 364
  6 months post-intervention | 64 | 51

3. Primary Outcome: Number of Participants Reporting Non-contact Sexual Violence
Description: Acts of non-contact sexual violence were assessed using 10 items from the Sexual Experiences Survey. The 10 items are scored on a scale from 0 (zero acts) to 3 (multiple acts), indicating how many times the participant reported engaging in an act. The numbers of participants indicating they engaged in at least one act of non-contact sexually violent behavior (scores of 1 or 2) in the past twelve months, for the baseline assessment, or since last completing the questionnaire are presented here.
Time Frame: Baseline, immediately after completing the 3 week intervention, 6 months after completing the intervention
Population: This analysis includes participants who completed the assessments at the indicated time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Health Education Control Condition | RealConsent
Number analyzed (Participants) | 397 | 396
Participants
  Baseline | 90 | 99
  Immediately post-intervention: number analyzed (Participants) | 377 | 374
  Immediately post-intervention | 70 | 56
  6 months post-intervention: number analyzed (Participants) | 375 | 364
  6 months post-intervention | 65 | 55

4. Primary Outcome: Number of Participants Reporting Prosocial Bystander Behavior
Description: Participants were asked if they had engaged in any of four prosocial bystander behaviors in the past 12 months (or since the last time completing the questionnaire). Items are scored as 0 = never performed, 1 = performed once, 2 = performed more than once. The numbers of participants who report engaging in at least one of four prosocial bystander behaviors at least once are presented here.
Time Frame: Six months following baseline
Population: This analysis includes participants who completed the assessments at the indicated time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Health Education Control Condition | RealConsent
Number analyzed (Participants) | 397 | 396
Participants
  Baseline | 258 | 258
  6 months post-intervention: number analyzed (Participants) | 375 | 364
  6 months post-intervention | 170 | 203

5. Secondary Outcome: Knowledge of Legal Definitions of Assault and Rape Scale Score
Description: Knowledge of the law is assessed with 22 items where respondents indicate if they think the situations described are illegal (scored as 1), legal, but harmful (2), or not sexual violence (3), with example items including "Forcing a person to have oral sex" and "Pressuring someone to have sex." Items were re-coded such that responses indicating an accurate estimate or overestimate of the illegality and harms of sexual violence were coded as "1" and items indicating an underestimation as of the illegality and harms of sexual violence were coded as "0". Total scores range from 0 to 22 with higher scores indicating greater awareness of laws and consequences related to sexual violence.
Time Frame: Baseline, immediately after completing the 3 week intervention, 6 months after completing the intervention
Population: This analysis includes participants who completed the assessments at the indicated time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Health Education Control Condition | RealConsent
Number analyzed (Participants) | 397 | 396
score on a scale
  Baseline | 16.94 (3.72) | 17.02 (3.52)
  Immediately post-intervention: number analyzed (Participants) | 377 | 374
  Immediately post-intervention | 18.01 (4.31) | 18.86 (4.02)
  6 months post-intervention: number analyzed (Participants) | 375 | 364
  6 months post-intervention | 18.43 (4.51) | 18.58 (5.05)

6. Secondary Outcome: Knowledge of Informed Consent to Have Sex Score
Description: Knowledge of sexual consent is assessed with 15 items where respondents indicate how much they agree with each statement on a 5-point Likert scale of 1 to 5, where 1 = totally agree and 5 = totally disagree. This scale was adapted from fifteen items of the Sexual Consent Attitudes and Behaviors scale. Example items include "The need to ask for sexual consent DECREASES as the length of a dating relationship INCREASES" and "If your partner initiates sexual contact, it is okay to continue, even if she/he is drunk". Several items were reverse-coded to maintain common valence, and all response options were re-coded to range from 0-4. Total scores range from 0 to 60 where higher scores indicate greater knowledge about sexual consent.
Time Frame: Baseline, immediately after completing the 3 week intervention, 6 months after completing the intervention
Population: This analysis includes participants who completed the assessments at the indicated time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Health Education Control Condition | RealConsent
Number analyzed (Participants) | 397 | 396
score on a scale
  Baseline | 34.33 (5.31) | 35.05 (5.83)
  Immediately post-intervention: number analyzed (Participants) | 377 | 374
  Immediately post-intervention | 33.94 (6.06) | 35.81 (7.68)
  6 months post-intervention: number analyzed (Participants) | 375 | 364
  6 months post-intervention | 33.64 (6.51) | 35.54 (7.50)

7. Secondary Outcome: Gender Roles Score
Description: The Gender Role Attitudes (GRA) scale measures men's gender role attitudes. The fifteen-item scale was adapted from the Gender Equitable Men (GEM) scale, a scale that was adapted for use in Nepal from the GEM scale, the Male Role Norms Inventory (MRNI)-Adolescent-revised scale, the Gender Attitudes Scale, and the International Men and Gender Equality Survey (IMAGES). Example items included: "A woman should obey her husband even when she disagrees with him" and "Men should be the ones to initiate dating relationships". Response options were coded using a 5-point Likert scale ranging from totally agree (1) to totally disagree (5). Two items needed to be reverse coded to maintain common valence, and all items were re-coded to range from 0-4, resulting in a theoretical score range of 0-60, with higher scores indicating more equitable attitudes.
Time Frame: Baseline, immediately after completing the 3 week intervention, 6 months after completing the intervention
Population: This analysis includes participants who completed the assessments at the indicated time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Health Education Control Condition | RealConsent
Number analyzed (Participants) | 397 | 396
score on a scale
  Baseline | 38.34 (7.14) | 38.82 (7.53)
  Immediately post-intervention: number analyzed (Participants) | 377 | 374
  Immediately post-intervention | 36.15 (8.08) | 37.21 (9.10)
  6 months post-intervention: number analyzed (Participants) | 375 | 364
  6 months post-intervention | 35.43 (8.72) | 36.77 (9.61)

8. Secondary Outcome: Myths and Realities About Sexual Violence Score
Description: Beliefs about what other men think about myths and realities of sexual violence was to be assessed with 24 items asking respondents to indicate how much they agree with each statement. Responses were to be given on a scale from 1 to 5 where 1 = totally agree and 5 = totally disagree. Total scores range from 24 to 120 with lower scores indicating that the respondent thinks men his age agree more with myths concerning sexual violence.
Time Frame: Baseline, Posttest (immediately after completing the intervention), 6 Months after intervention
Population: Data for this outcome were not collected as the items performed poorly during pilot testing and this questionnaire was not administered to study participants.
Arm/Group | Health Education Control Condition | RealConsent
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Sexual Coercion Score
Description: This 19-item scale was adapted from the Sexual Coercion in Intimate Relationships scale. Examples of items in the scale included: "Saying that a person would have sex with you if they truly love you" and "Asking your dating partner repeatedly to perform a sexual act after they have said that they do not want to". Response options were coded into "No" (0), "Yes" (1) and "Unsure" (2). Three items had to be reverse coded to maintain common valence. For analysis, "No" and "Unsure" were re-coded into one response option. Scores range from 0-19. Higher scores indicate a greater understanding of behaviors that are sexually coercive.
Time Frame: Baseline, Posttest (immediately after completing the intervention), 6 Months after intervention
Population: This analysis includes participants who completed the assessments at the indicated time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Health Education Control Condition | RealConsent
Number analyzed (Participants) | 397 | 396
score on a scale
  Baseline | 5.74 (5.59) | 5.76 (5.69)
  Immediately post-intervention: number analyzed (Participants) | 377 | 374
  Immediately post-intervention | 5.61 (5.71) | 6.45 (6.39)
  6 months post-intervention: number analyzed (Participants) | 375 | 364
  6 months post-intervention | 5.54 (5.74) | 5.90 (6.18)

10. Secondary Outcome: Sexual Violence Myths Score
Description: Rape attitudes were assessed with 28 items presenting myths about rape. Items are scored on a 5-point Likert scale from 1 to 5 where 1 = totally agree and 5 = totally disagree. The Rape Myth Attitudes (RMA) scale measures the extent of men's endorsement (or non-endorsement) of common rape myths. This scale was adapted from fourteen items of the Illinois Rape Myth Scale-Short Form and eleven items of the College Date Rape Attitude and Behavior Survey. Example items included: "When guys rape, it is usually because of their strong desire for sex" and "In most cases when a woman was raped, she was asking for it". Several items were reverse-coded to maintain common valence, and all response options were re-coded 0-4, resulting in a theoretical range of 0-112, with higher scores indicating less endorsement of rape myths.
Time Frame: Baseline, immediately after completing the 3 week intervention, 6 months after completing the intervention
Population: This analysis includes participants who completed the assessments at the indicated time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Health Education Control Condition | RealConsent
Number analyzed (Participants) | 397 | 396
score on a scale
  Baseline | 40.38 (7.83) | 40.89 (8.47)
  Immediately post-intervention: number analyzed (Participants) | 377 | 374
  Immediately post-intervention | 39.95 (9.02) | 43.01 (11.37)
  6 months post-intervention: number analyzed (Participants) | 375 | 364
  6 months post-intervention | 41.61 (10.13) | 44.34 (12.68)

11. Secondary Outcome: Alcohol and Consent Score
Description: Beliefs about consent in terms of alcohol use are assessed with 5 items adapted from the College Date Rape Attitudes and Behaviors scale where respondents indicate how much they agree with each statement. Responses are on a scale from 1 = totally agree to 5 = totally disagree. Items were re-coded to be grounded at zero. Total scores range from 0 to 20 where higher scores indicate more understanding of sexual consent under the influence of alcohol.
Time Frame: Baseline, immediately after completing the 3 week intervention, 6 months after completing the intervention
Population: This analysis includes participants who completed the assessments at the indicated time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Health Education Control Condition | RealConsent
Number analyzed (Participants) | 397 | 396
score on a scale
  Baseline | 14.57 (2.88) | 15.04 (2.95)
  Immediately post-intervention: number analyzed (Participants) | 377 | 374
  Immediately post-intervention | 14.18 (2.77) | 15.45 (3.38)
  6 months post-intervention: number analyzed (Participants) | 375 | 364
  6 months post-intervention | 14.30 (2.91) | 15.06 (3.52)

12. Secondary Outcome: Rape Empathy Score
Description: Empathy for rape victims was assessed with a modified version of the Rape Empathy Scale (RES). This assessment includes 17 items where participants were asked to choose between two statements, one of which reflected greater empathy towards rapists ("I understand the helplessness a rapist might feel during a rape, since he cannot control his actions") and one of which reflected greater empathy towards victims ("I understand the helplessness a victim might feel during a rape"). Responses are scored as 1 (more empathy for victim) or 0 (more empathy for perpetrator) and total scores range from 0 to 17 where higher scores indicate more empathy towards rape victims.
Time Frame: Baseline, immediately after completing the 3 week intervention, 6 months after completing the intervention
Population: This analysis includes participants who completed the assessments at the indicated time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Health Education Control Condition | RealConsent
Number analyzed (Participants) | 397 | 396
score on a scale
  Baseline | 11.61 (2.66) | 11.46 (2.73)
  Immediately post-intervention: number analyzed (Participants) | 377 | 374
  Immediately post-intervention | 11.41 (2.99) | 12.01 (3.27)
  6 months post-intervention: number analyzed (Participants) | 375 | 364
  6 months post-intervention | 11.64 (3.17) | 11.97 (3.47)

ADVERSE EVENTS:
Time Frame: Information on adverse events was collected from participants for 14 months.
Arm/Group | Health Education Control Condition | RealConsent
All-Cause Mortality (participants affected / at risk) | 0/397 | 0/396
Serious Adverse Events (participants affected / at risk) | 0/397 | 0/396
Other Adverse Events (participants affected / at risk) | 0/397 | 0/396

LIMITATIONS AND CAVEATS:
The 12-month follow-up period allowed for a short-term impact assessment of the intervention. Longer-term follow-up of participants is needed to assess the impact of the intervention on behavioral outcomes throughout men's time at university, and beyond.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-16): https://cdn.clinicaltrials.gov/large-docs/55/NCT04147455/Prot_SAP_001.pdf